CLINICAL TRIAL: NCT06878443
Title: Multicentric Clinical Pilot Essay Testing Association Between Antibiotics and Vaginal Probiotics for Patients With Prematured Rupture of Membranes Between 32 and 36 Weeks of Amenorrhea ( PROBPROM-Pilot Study)
Brief Title: Vaginal Probiotics During Pregnancy After Premature Rupture of Membranes
Acronym: PROBPROM-Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Important delays limiting study starts
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-02-2025-12298
Record Dates: First submitted 2024-09-10; First posted 2025-03-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy; Prematurity; PPROM
Keywords: pregnancy; prematurity; PPROM; vaginal probiotics; microbiota
MeSH Terms: conditions — Premature Birth; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Intervention Model Description: Vaginal Probiotics 1x/day until delivery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotics group (Experimental): Pregnant women admitted to one of the center participating in the essay for PPROM accepting vaginal probiotics intake and sample collection
  Interventions: Other: Vaginal probiotics
- Control group - PPROM (No Intervention): Pregnant women admitted to one of the study's centers for PPROM without vaginal probiotics intake
- Control group- Full Term (No Intervention): Pregnant women with expected full-term deliveries, without vaginal probiotics intake

INTERVENTIONS:
Other: Vaginal probiotics — Probiotics from Canadian company Lallemand Health Solutions are stored at room temperature and administered vaginally.
  Arms: Probiotics group

SUMMARY:
The goal of this clinical trial is to compare the microbiota of preterm babies born after premature breaking water with full-term babies microbiota.

The main questions it aims to answer are:

* Is babies' microbiota differs with premature water breaking than full-term babies microbiota?
* Is vaginal probiotics given to the mother influence the baby microbiota? Researchers will compare vaginal probiotics use to no treatment to see if the babies microbiota and mother microbiota is influenced.

Participants will

* Take vaginal probiotics between premature breaking water until delivery (group A)
* Keep a diary of their symptoms and compliance to treatment (group A)
* Take samples of vaginal secretions and of baby's stool (all groups)

DETAILED DESCRIPTION:
Premature rupture of fetal membranes before labor (PPROM) reprensents 30% of premature births. As PPROM is strongly associated with ascending vaginal infection, antibiotics are recommended during the latent period (LP) (the interval between rupture and birth). They prolong the LP and improve the health of the children, but they also aggravate pre-existing vaginal dysbiosis. The addition of vaginal probiotics (VP) stabilizes the vaginal microbiota (VM) and increases Lactobacillus levels. By increasing the number of good germs in the vagina, they will rebalance the good germs and the pathogenic germs that make their way up to the uterus. This could reduce uterine infection and improve the foetus; intestinal flora.

Pathophysiological hypotheses for improving neonatal health:

The use of VP could have three modes of action on neonatal outcome:

i) decrease vaginal dysbiosis: pregnancy prolongation and reduce fetal immaturity complications (e.g.reduce intraventricular hemorrhage); ii) Reduction of intra-uterine infection/inflammation: Reduce neonatal complications linked to inflammation (e.g. diminish cystic periventricular leukomalacia); iii) improvement of neonatal intestinal microbiota (NIM) (probiotic swallowing): reduce complications associated with neonatal dysbiosis (e.g. reduce ulcerative colitis (NEC)).

3.1 Primary objective Mechanistic proof of concept To compare the NIM of the babies of the participants after PPROM with or without probiotics compared with the NIM of the babies of the participants without PRPOM (meconium and at 7 days of life).

Secondary objectives Primary secondary objectives (Group A or B versus C)

1. To compare the VM of participants after PPROM with or without probiotics with the VM of participants without PPROM at the end of pregnancy (early latency phase).
2. Compare the VM of participants after PPROM with or without probiotics with the VM of participants without PPROM in early labor (end of latency phase).
3. To test the possibility of transmission analysis of VP in the NIM (meconium and at 7 d of life) with groups B and C: PPROM-control and control without PPROM.

Secondary clinical objectives

1. Explore recruitment (rate, reasons for acceptance and refusal, characteristics of mothers recruited), treatment adherence >80% and attrition rate <5%.
2. Test tools for sample collection, participant information and consent form.

Population:

Pregnant women aged 18 and over, giving birth at one the three centers participating in the study CHUM, CHUSJ or CHUQ (Quebec). These women will be divided into 3 groups:

* Group A: PPROM-VP Pregnant women admitted for PPROM with VP intake
* Group B: PPROM-control Pregnant women admitted for PPROM without VP intake
* Group C: term-control without PPROM Pregnant women with expected full-term deliveries, without VP intake

ELIGIBILITY:
Inclusion Criteria:

* Groups A and B:

Women ≥ 18 years of age, mono-fetal pregnancy, hospitalized for PPROM between 32 0/7 d and 36 0/7 d weeks of ammenorhea with LP < 7 days in one of the participating centers, with expectant management, who have consented to participate, agree to collect samples and speak French or English

Group C:

Women ≥ 18 years, mono-fetal pregnancy, expected delivery in one of the participating centers and speaking French or English

Exclusion Criteria:

* Groups A and B:
* Presence of active labor,
* Situations contraindicating expectant management (e.g. infection),
* Significant malformation, chromosomal abnormality or fetal death,
* Signs of fetal distress,
* vaginal probiotics intake 15 days before study entry.

For Group A only:

* Allergies to soy and/or milk;
* Weakened immune system (e.g. AIDS, prolonged treatment with corticosteroids),
* Not to have been treated with the following antibiotics during pregnancy: nalidixic acid (Negram) and/or cefoxitin (Mefoxin) and/or sulfamethoxazole (Bactrim).

Group C:

* History of obstetric complications (prematurity <37 weeks, diagnosed pre-eclampsia, gestational diabetes treated with insulin),
* Known obstetrical or fetal complications of the current pregnancy, such as threat of preterm delivery (premature rupture of membranes or preterm labor), chorioamnionitis, placenta previa, active vaginal bleeding, cervical cerclage, fetal distress or malformation, corticosteroid therapy,
* Risk factors for obstetrical complications during pregnancy, such as gestational diabetes, type I/II diabetes and high blood pressure (systole ≥ 140 and diastole ≥ 90),
* Antibiotics taken 15 days prior to inclusion,
* Taking probiotics 15 days prior to inclusion,
* Tested positive for Streptococcus group B during previous pregnancies (as this will require antibiotics at delivery),
* Presence of symptoms such as fever, nausea, vomiting, bloody diarrhea or severe abdominal pain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Probiotics primers presence | at birth and 7th day of life
  Evaluate the presence or absence of probiotics in the meconium and stools of 7-day-old babies using specific primers to detect strains

SECONDARY OUTCOMES:
Recruitment rate | 12 months
  To assess feasability of the study the recruitment will be explored (recruitment rate = (# of eligible patient- # of patient who didn't consent) / # of eligible patient), also, reasons for acceptance and refusal, characteristics of mothers recruited will be documented.
Numbers of mother and baby health issues | During the enrollment until 30 days after delivery
  Monitor side-effects reported in the logbook and medical record, as well as clinical outcomes for mother and baby
Probiotics primers in other samples presence | between the enrollment until 30 days after delivery
  Evaluate the presence or absence of probiotics in the various samples, i.e. vaginal secretions, meconium and 7-day-old baby's stools, using specific primers to detect strains, and ii) perform microbiota analysis to compare the microbiota of mothers with and without PPROM.
Attrition rate | 13 months
  To assess feasability of the study, the attrition rate will be explored. Attrititon rate = (# participants who dropped out / total of participants)
Treatment adherence | 13 months
  # of caps took during the treatment phase will be reported to explore the adherence of treatment. This will help to assess feasability of the study

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM Clinical research Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided